CLINICAL TRIAL: NCT05060367
Title: Pharmacokinetic Analysis of Nutrient Absorption From a Novel Liposomal Multivitamin/Mineral Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Nutraceutical Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2021-527
Record Dates: First submitted 2021-09-10; First posted 2021-09-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Mineral Absorption
MeSH Terms: interventions — Minerals

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal multivitamin/mineral condition (Experimental): Ingestion of novel, liposomal multivitamin/mineral.
  Interventions: Dietary Supplement: Liposomal multivitamin/mineral
- Standard multivitamin/mineral condition (Active Comparator): Ingestion of standard multivitamin/mineral.
  Interventions: Dietary Supplement: Standard multivitamin/mineral

INTERVENTIONS:
Dietary Supplement: Liposomal multivitamin/mineral — Two-capsule dose of liposomal multivitamin/mineral that is nutrient-matched to the standard multivitamin/mineral.
  Arms: Liposomal multivitamin/mineral condition
Dietary Supplement: Standard multivitamin/mineral — Two-capsule dose of standard multivitamin/mineral that is nutrient-matched to the liposomal multivitamin/mineral.
  Arms: Standard multivitamin/mineral condition

SUMMARY:
This project is a randomized crossover trial examining the pharmacokinetic profiles of standard and liposomal multivitamin/mineral (MVM) formulations in healthy adults. Each participant will complete two research visits, which will be identical except for which MVM product is consumed. At each visit, participants will report to the laboratory after an overnight fast. After a baseline blood sample is collected, the MVM product will be consumed alongside a standardized breakfast. At 2-, 4-, and 6-hours post-ingestion, additional blood samples will be collected. Concentrations of representative minerals will be analyzed to determine whether differential nutrient absorption is observed with the liposomal MVM as compared to the standard MVM product. The results of this study will provide information about a novel liposomal MVM formulation and will inform future research and commercial applications of this technology.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65 at time of consent
2. ability to comply with study procedures
3. availability to complete study based on durations of individual visits and scheduling requirements
4. body mass of at least 110 pounds

Exclusion Criteria:

1. failure to meet any of the aforementioned inclusion criteria
2. presence of a disease or medical condition that could reasonably influence study outcomes or make participation inadvisable
3. use of medication that could reasonably influence study outcomes or make participation inadvisable
4. inability to abstain from medication, supplement, or substance use during the overnight fast and duration of the study visit
5. anticipated inability to provide blood samples (e.g., known difficulty providing blood samples)
6. currently pregnant or breastfeeding, based on self-report
7. allergy that would prevent safe consumption of standardized breakfast or multivitamin product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Iron | The AUC value will be calculated using data from four time points: immediately prior to multivitamin/mineral ingestion and 2, 4, and 6 hours after ingestion of multivitamin/mineral.
  Area under the concentration vs. time curve (AUC) for iron in serum
Iron | The Cmax value will be determined as the highest concentration observed from four time points: immediately prior to multivitamin/mineral ingestion and 2, 4, and 6 hours after ingestion of multivitamin/mineral.
  Maximal concentration (Cmax) of iron in serum
Magnesium | The AUC value will be calculated using data from four time points: immediately prior to multivitamin/mineral ingestion and 2, 4, and 6 hours after ingestion of multivitamin/mineral.
  Area under the concentration vs. time curve (AUC) for magnesium in serum
Magnesium | The Cmax value will be determined as the highest concentration observed from four time points: immediately prior to multivitamin/mineral ingestion and 2, 4, and 6 hours after ingestion of multivitamin/mineral.
  Maximal concentration (Cmax) of magnesium in serum

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No